CLINICAL TRIAL: NCT03883841
Title: Fetal Vascular Hemodynamic Changes Before and After Treatment of Maternal Iron Deficiency Anemia
Brief Title: Fetal Vascular Hemodynamic Changes in Iron Deficiency Anemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: DIDA
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Injections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: patients with iron deficiency anemia
  Interventions: Drug: Iron Sucrose Solution for Injection
- control group: normal pregnant patients

INTERVENTIONS:
Drug: Iron Sucrose Solution for Injection — intravenous infusion of iron sucrose
  Groups: Study group

SUMMARY:
Iron deficiency anemia is a worldwide medical disorder. So far, it is the most common medical complication in pregnancy specially in developing countries. It is the cause of many adverse effects on mother and fetus and contributes significantly to high maternal mortality. Maternal iron deficiency anemia is frequently associated with premature delivery, low birth weight babies

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational age 28-32 weeks
* singleton pregnancy
* iron deficiency anemia.

Exclusion Criteria:

* Multiple pregnancy
* antepartum hemorrhage
* major congenital fetal anomalies
* any other type of anemia other than iron deficiency anemia
* any acute or chronic maternal disease other than iron deficiency anemia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes pregnant women 28 - 32 week gestation (calculated by the last menstrual period or by earlier ultrasound examination)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The mean changes in middle cerebral artery Doppler of the fetus | one month
  Doppler evaluation